CLINICAL TRIAL: NCT06308380
Title: Effectiveness of Rehabilitation Protocol in Patients With Shortened Posterior Leg Muscles, Whether or Not Combined With Ultrasound- Guided Surgery
Brief Title: Effectiveness of Rehabilitation Protocol in Patients With Shortened Posterior Leg Muscles
Acronym: EREPSOLM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCV/2022-2023/158
Record Dates: First submitted 2024-01-19; First posted 2024-03-13 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-07

CONDITIONS: Equinus Deformity of Foot; Gastrocnemius Equinus; Contracture
Keywords: foot deformity; calf shortening; foot and ankle disease; stretching and muscle strengthening; exercise post surgery
MeSH Terms: conditions — Contracture; Foot Deformities | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rehabilitation only (Active Comparator): All patients who do not wish to undergo mini- invasive surgery to lengthen the calf muscles are part of the control group. They will be subjected to a specific protocol of rehabilitation exercise 3times a week for 12 weeks.
  Interventions: Procedure: Specific protocol of rehabilitation exercise
- Surgery (Experimental): All patients who wish to undergo mini invasive surgery to lengthen the calf muscles are part of the experimental group. they will be subjected to a specific protocol of rehabilitation exercise exercise 3times a day every day for 4weeks.
  Interventions: Procedure: Specific protocol of rehabilitation exercise; Procedure: Short gastrocnemius surgery.

INTERVENTIONS:
Procedure: Specific protocol of rehabilitation exercise — Specific protocol of rehabilitation exercise
  Other Names: Exercise
Procedure: Short gastrocnemius surgery. — During surgery, a partial release of the gastrocnemius muscle tendon is performed to relieve tension and allow greater range of motion. This procedure is typically performed on an outpatient basis and under local or regional anesthesia, which allows for a quicker recovery compared to more invasive surgeries.
  Arms: Surgery

SUMMARY:
The goal of this clinical study is to develop a specialized rehabilitation exercise protocol designed for patients diagnosed with foot pathologies and calf muscle shortening, regardless of their choice to undergo minimally invasive ultrasound-guided surgery. The primary focus is to assess disparities in outcomes, particularly in the recovery of ankle mobility degrees. Additionally, for patients opting for minimally invasive ultrasound-guided surgery, the study aims to evaluate the resumption of both sporting activities and daily routines using the aforementioned specific rehabilitation protocol.

The primary questions this study aims to answer are:

* How does the proposed rehabilitation protocol impact ankle mobility recovery for patients with foot pathologies and calf muscle shortening?
* What are the differences observed in the return to sporting activities and daily life among patients undergoing minimally invasive ultrasound-guided surgery, following the prescribed protocol?

Participants enrolled in this study will be engaged in:

Undertaking the specified rehabilitation exercises tailored for foot pathologies and calf muscle shortening.

Those opting for minimally invasive ultrasound-guided surgery will follow the same rehabilitation protocol post-surgery to assess its impact on their return to normal activities.

If there exists a comparison group:

Researchers will compare participants who undergo minimally invasive ultrasound-guided surgery against those who choose other treatment options to discern any differential effects on ankle mobility recovery and resumption of activities.

DETAILED DESCRIPTION:
Calf muscle tightness and limited ankle dorsiflexion range of motion are associated with various foot pathologies, including plantar fasciitis, Achilles tendinitis, and altered gait patterns. While conservative rehabilitation exercises are first-line treatment, minimally invasive ultrasound-guided gastrocnemius recession can be considered for refractory cases. However, no studies have compared using the same rehabilitation protocol post-surgery versus without surgery. The aim of this randomized controlled trial is to evaluate the efficacy of a specialized 12-week rehabilitation protocol on ankle dorsiflexion range of motion in patients with foot pathologies and calf tightness. Secondary objectives are to compare post-surgical outcomes in patients undergoing minimally invasive ultrasound-guided gastrocnemius recession followed by the 12-week rehabilitation protocol, versus patients only undergoing the rehabilitation protocol, in terms of ankle dorsiflexion range of motion, foot posture and plantar pressures, pain scores, function scores, and return to activities.

A parallel group design will be used, with participants assigned to two groups: Group A will undergo the rehabilitation protocol only and Group B will undergo the rehabilitation protocol after ultrasound-assisted gastrocnemius surgery. Adult patients between 20 and 90 years of age with clubfoot pathology and gastrocsoleus contracture with calf strain will be recruited. The target sample size is 40 patients, equally distributed in the two groups.

The study protocol will consist of assessing participants at baseline for calf muscle length, ankle dorsiflexion range of motion, foot posture, plantar pressures, pain and function. Group A will undergo the 12-week rehabilitation protocol. Group B will undergo ultrasound-guided minimally invasive surgery first, followed by the 12-week rehabilitation protocol. Evaluations will be performed at Pre-surgery, 2 months, 6 months.

Statistical analysis will compare the two groups on all outcome measures using appropriate statistical tests. Expected results are improved ankle dorsiflexion range of motion in both groups, with greater improvements in Group B post-surgery. This study will provide evidence on a targeted rehabilitation protocol for calf tightness, and also insight into the added benefits of minimally invasive surgery when combined with focused rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with shortened posterior musculature.
* Chronic ankle pain.
* Limitations in activities of daily living.
* Atypical gait.
* Clubfoot.

Exclusion Criteria:

* Previous MMII surgeries.
* Neuropathic pain.
* Bony cap equinus.
* Analgesic physiotherapy.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Gait Analysis | Pre-surgery, 2 months, 6 months.
  The Gait Analysis is an examination useful for studying patterns, aided by instruments that measure the load on each limb and overall ambulation. The gait cycle ia s particularly complex phenomenon, resulting from the coordination between the nervous system, musculoskeletal system, and sensory input. The patient is required to walk (at varying intervals) on a treadmill or directly on a platform. It's a non invasive examination.
Baropodometric examination | Pre-surgery, 2 months, 6 months.
  The baropodometric examination, a pivotal tool in studying plantar pressure distribution, is conducted on the Zebris platform. This platform provides a detailed and precise analysis of pressures exerted on the plantar surface during walking, enabling a comprehensive assessment of alterations in load distribution on the feet. Zebris' technology allows for gathering relevant data on pressure points and load areas, facilitating the identification of abnormal gait patterns and postural imbalances. Integrated within the Zebris platform, this examination becomes an invaluable resource for comprehensive biomechanical assessment and personalized treatment planning for various foot pathologies.

SECONDARY OUTCOMES:
Passive ankle mobility | Pre-surgery, 2 months, 6 months.
  It is a tool that measures muscle strength and is used to evaluate the Passive ankle mobility test. The latter allows us to evaluate the equine.Measurement in degrees.
Short Form Health Survey 36 score | Pre-surgery, 2 months, 6 months.
  It's a self administered questionnaire filled out by the patient, aimed at quantifying health status and measuring health related quality of life.
  On this 0 - 100 scale of the The Short Form-36 Health Survey(SF-36), the higher the score obtained, the better the health status. Thus, 0 represents the worst state of health and 100 the best state of health as measured by the SF-36.
Foot Function Index | Pre-surgery, 2 months, 6 months.
  It is a questionnaire consisting of 23 items designed to assess the impact that foot pathologies have on the patient's perceived health status in terms of pain, disability and activity limitation.
American Orthopedic Foot and Ankle Score | Pre-surgery, 2 months, 6 months.
  The AOFAS Ankle-Hindfoot Scale was designed by the American Foot and Ankle Society to provide an international method to assess the clinical status of the ankle and foot.
  This questionnaire incorporates subjective and objective factors that are scored using a numerical scale and describe variables of function, alignment and pain. The score ranges from 0 to 100 depending on the degree of limitation of the patient.
Halasi score | Pre-surgery, 2 months, 6 months.
  The Halasi Ankle Activity Score is a ten-point scoring system in which various sports and physical activities are divided into 10 groups according to the biomechanical load on the ankle; for each sport discipline, three levels can be selected ranging from recreational level (more than one hour per week) to professional or international elite level.

OTHER OUTCOMES:
Olerud and Molander ankle score. | Pre-surgery, 2 months, 6 months.
  it is a functional assessment scale that uses a numerical scoring approach to measure a patient's function or status in relation to nine different items. In this case, the variable measured through this scale is a continuous quantitative variable. the scale assigns scores ranging from 0 to 100, based on the patient's responses or evaluations regarding the nine mentioned items. Higher scores indicate better functioning or a more favorable health status, while lower scores indicate impaired functioning or a less favorable health state.
Visual Analogue Scale | Pre-surgery, 2 months, 6 months.
  A 10-centimeter horizontal line is used, with extreme expressions of a symptom at both ends; absence or lesser intensity on the left and greater intensity on the right. The patient marks the point indicating intensity, measures it with a millimeter ruler, and expresses it in centimeters. The classification is: Mild pain (less than 3), moderate pain (between 4 and 7), and severe pain (8 or higher).

CONTACTS AND LOCATIONS:
Overall Officials: Javier Ferrer-Torregrosa, Dr., Study Director — FundaciónUcv; Juan Vicente-Mampel, Dr., Study Director — FundaciónUcv
Locations (3):
- Spain (3):
  - Podologia Avançada, Granollers, Barcelona
  - Clinica Mayral foot center, Barcelona, Barcelon
  - Clinicas UCV, Valencia, València

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pearce CJ, Seow D, Lau BP. Correlation Between Gastrocnemius Tightness and Heel Pain Severity in Plantar Fasciitis. Foot Ankle Int. 2021 Jan;42(1):76-82. doi: 10.1177/1071100720955144. Epub 2020 Sep 13. PMID 32924578
- [Background] Nakale NT, Strydom A, Saragas NP, Ferrao PNF. Association Between Plantar Fasciitis and Isolated Gastrocnemius Tightness. Foot Ankle Int. 2018 Mar;39(3):271-277. doi: 10.1177/1071100717744175. Epub 2017 Dec 4. PMID 29198141
- [Background] Medeiros DM, Martini TF. Chronic effect of different types of stretching on ankle dorsiflexion range of motion: Systematic review and meta-analysis. Foot (Edinb). 2018 Mar;34:28-35. doi: 10.1016/j.foot.2017.09.006. Epub 2017 Oct 27. PMID 29223884
- [Background] Meyer DC, Werner CM, Wyss T, Vienne P. A mechanical equinometer to measure the range of motion of the ankle joint: interobserver and intraobserver reliability. Foot Ankle Int. 2006 Mar;27(3):202-5. doi: 10.1177/107110070602700309. PMID 16539903
- [Background] Barouk P, Barouk LS. Clinical diagnosis of gastrocnemius tightness. Foot Ankle Clin. 2014 Dec;19(4):659-67. doi: 10.1016/j.fcl.2014.08.004. Epub 2014 Sep 26. PMID 25456715
- [Background] Villanueva M, Iborra A, Rodriguez G, Sanz-Ruiz P. Ultrasound-guided gastrocnemius recession: a new ultra-minimally invasive surgical technique. BMC Musculoskelet Disord. 2016 Oct 3;17(1):409. doi: 10.1186/s12891-016-1265-7. PMID 27716217
- [Background] Moroni S, Fernandez-Gibello A, Nieves GC, Montes R, Zwierzina M, Vazquez T, Garcia-Escudero M, Duparc F, Moriggl B, Konschake M. Anatomical basis of a safe mini-invasive technique for lengthening of the anterior gastrocnemius aponeurosis. Surg Radiol Anat. 2021 Jan;43(1):53-61. doi: 10.1007/s00276-020-02536-1. Epub 2020 Jul 23. PMID 32705404
- [Background] Baraja-Vegas L, Martin-Rodriguez S, Piqueras-Sanchiz F, Faundez-Aguilera J, Bautista IJ, Barrios C, Garcia-Escudero M, Fernandez-de-Las-Penas C. Localization of Muscle Edema and Changes on Muscle Contractility After Dry Needling of Latent Trigger Points in the Gastrocnemius Muscle. Pain Med. 2019 Jul 1;20(7):1387-1394. doi: 10.1093/pm/pny306. PMID 30715456
- [Background] Cobacho MT, Barcia JM, Freijo-Gutierrez V, Caballero-Gomez F, Ferrer-Torregrosa J. A Predictive Model for Gastrocnemius Tightness in Forefoot Pain and Intractable Plantar Keratosis of the Second Rocker. J Am Podiatr Med Assoc. 2021 May 1;111(3):Article_12. doi: 10.7547/18-024. PMID 34144595
- [Background] Head J, Mallows A, Debenham J, Travers MJ, Allen L. The efficacy of loading programmes for improving patient-reported outcomes in chronic midportion Achilles tendinopathy: A systematic review. Musculoskeletal Care. 2019 Dec;17(4):283-299. doi: 10.1002/msc.1428. Epub 2019 Nov 25. PMID 31763774